CLINICAL TRIAL: NCT01816542
Title: Dermatologically Tested - Patch Tests - to Assess the Irritancy/Allergic Sensitivity of the Natural Personal-care Products Developed by "Mother's Choice".
Brief Title: Evaluation of Irritancy/Allergic Sensitivity to Natural Personal-care Products by Patch Tests
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mother's Choice Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MC-2013-PT-BA
Record Dates: First submitted 2013-02-12; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Cutaneous Patch; Dermatitis; Allergy; Cosmetic Allergy; Eczema; Contact, Allergic
Keywords: patch-testing; personal-care; cosmetic; dermatitis; allergy; sensitive skin
MeSH Terms: conditions — Plaque, Amyloid; Dermatitis; Hypersensitivity; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patch tests on healthy skin (Other)
  Interventions: Other: patch tests on healthy skin

INTERVENTIONS:
Other: patch tests on healthy skin — Patches will be placed on healthy skin.

SUMMARY:
The purpose of the study is to determine if any of Mother's Choice' all-natural personal-care products cause either irritation or allergic reaction when applied to both normal or sensitive skin.

Each product will be tested on the skin using patch tests.

DETAILED DESCRIPTION:
Volunteers will be seen on Day #0 and the study purpose will be explained. Each volunteer will be interviewed to determine if he/she has any exclusion criteria.

If there is no contraindication, and agreement is achieved,consent forms will be signed.

Volunteers will be examined by a lactic acid test to determine if he/she has normal or sensitive skin. In this test, a Finn's cell (plastic cell, size 1*1 cm) with lactic acid (50 microliter, 10%w/v) will be placed on the volunteer's cheek for ten minutes. The volunteer will be defined as "sensitive" or "normal" according to the degree of discomfort they report.

Patch-tests will be performed in the standard method. The materials to be tested will be placed in Finn's cells and attached to the participants healthy skin's back by a plaster (Micropore).The chambers will be left on the skin for 48 hours. The test will be read by a specialist one hour after chambers' removal and 48 hours afterwards. Any erythema,edema, blisters, pustules or erosions on the skin in the patch area will be considered a positive response, and will be evaluated by clinical tools as being of the irritant or the allergic type. in case of uncertainty we may use a confocal microscope for in vivo diagnosis.

Ingredients: appropriate concentrations and solvents of the test materials will be prepared according to accepted standards (refer to: Anton C. De Groot: Patch Testing, 3ed Edition, Wapserveen, The Netherlands, 2009).Leave on products will be tested 'as is'. Rinse off products will be diluted to 5% and 0.5%.

If the skin stays normal after the patch removal, it means that contact with the material did not cause allergy or irritation.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adults

Exclusion Criteria:

* Pregnant subjects
* Subjects with an allergy or a skin disease which interferes with the proper results of the tests.
* Subjects who are taking medications which can interfere with the proper results of the tests. For example: systemic corticosteroids, topical steroids applied to the test area.
* Subjects with sun or phototherapy induced tanning at the test area.
* Subject who had been participating in allergy tests within eight weeks prior to the present tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with positive reactions, number of positive reactions. | One week
  Erythema, edema, blisters, pustules or erosions on the skin in the patch area will be considered a positive response.
  If the skin is normal after the patch removal, it means that contact with the material do not cause allergy or irritation.

SECONDARY OUTCOMES:
Number of irritant versus allergic reactions, as determined by confocal microscopy. | On the spot
  In case of a positive reaction, it will be examined by confocal microscopy, by a specialist, to determine whether the reaction is irritant or allergic in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Ingber, MD Prof., Principal Investigator — Hadassah University Hospital, Department of Dermatology; Liran Horev, MD, Principal Investigator — Hadassah University Hospital, Department of Dermatology
Locations (1):
- Department of Dermatology, Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Mahmood T, Akhtar N. Short term study of human skin irritation by single application closed patch test: assessment of four multiple emulsion formulations loaded with botanical extracts. Cutan Ocul Toxicol. 2013 Mar;32(1):35-40. doi: 10.3109/15569527.2012.700472. Epub 2012 Jul 5. PMID 22765292
- [Background] Davies RF, Johnston GA. New and emerging cosmetic allergens. Clin Dermatol. 2011 May-Jun;29(3):311-5. doi: 10.1016/j.clindermatol.2010.11.010. PMID 21496740